CLINICAL TRIAL: NCT01686854
Title: "Terapia Dell'obesità: Studio Randomizzato Per la Valutazione Dell'Efficacia Della Terapia Cognitivo-comportamentale Versus Dietoterapia Prescrittiva Nel Controllo a Breve e Medio Termine Del Peso Corporeo e Del Rischio Cardiovascolare."
Brief Title: Effectiveness of Cognitive Behavioral Therapy vs. Prescriptive Diet in Short and Medium-term Control of Body Weight
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Chiara Muggia, dirigente medico 1° livello, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PSMCM01
Record Dates: First submitted 2012-05-29; First posted 2012-09-18 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Obesity
Keywords: cognitive-behavioral approach; obesity treatment
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral (B) (Experimental): a 12 months training program in small groups (max 10 persons) about problem solving strategies. Each 90 minute lesson will be given by clinicians, psicologist, dieticians, according cognitive behavioural approach and strategies.
  Interventions: Behavioral: Cognitive Behavioral (B)
- Prescriptive Diet (A) (Active Comparator): prescribed diet, with a reduction of 500 Kcal for overweight-1° degree obese, and of 800-1000 Kcal for 2° degree obese patients respect caloric requirement, in compliance with Italian guidelines (INRAN 2003).
  Interventions: Other: Prescriptive Diet (A)

INTERVENTIONS:
Behavioral: Cognitive Behavioral (B) — a 12 months training program in small groups (max 10 persons) about problem solving strategies. Each 90 minute lesson will be given by clinicians, psicologist, dieticians, according cognitive behavioural approach and strategies.
  Arms: Cognitive Behavioral (B)
Other: Prescriptive Diet (A) — prescribed diet, with a reduction of 500 Kcal for overweight-1° degree obese, and of 800-1000 Kcal for 2° degree obese patients respect caloric requirement, in compliance with Italian guidelines (INRAN 2003).
  Arms: Prescriptive Diet (A)

SUMMARY:
Comparison between different treatments of obesity in the short and medium term: prescriptive diet therapy compared to to cognitive-behavioral approach in the treatment of obesity according to the method of clinical trial.

According to the Italian guidelines on obesity, the target to reach is the weight loss of 10% compared to the initial weight, obtained in six months and maintained for the next 5 years.

The guideline considers six months as the time required to lose weight, but many patients are not able to achieve this result. Since in clinical practice many patients fail to achieve this weight loss in six months, it was decided to extend to 12 months the time to reach the target. As an intermediate goal it has been proposed to achieve a weight loss of at least 5% on respect of the basal weight in six months.

DETAILED DESCRIPTION:
The hypotheses to be tested is that the addition of a short CBT, as it can be applied in a public outpatients, is able to improve the percentage of responders and to raise the proportion of subjects able to maintain the result over time.

ELIGIBILITY:
Inclusion Criteria:

Subjects with severe overweight (BMI 27-29.9) or obesity of first step (BMI 30-34.9kg/h2 and obesity of second step (BMI 35-39.9 9kg/h2). Patients with dyslipidemia, hypertension, slight organ damage were eligible in the study; Exclusion Criteria:

patients treated with anorectic, estrogen or progestin and patients with diabetes or eating disordes were excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2007-03; Primary Completion 2012-01 (Actual); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
body weight reduction by 10% compared to the initial weight to over 12 months achievement of weight loss corresponding to 10% of the initial weight | 12 months
  body weight reduction by 10% compared to the initial weight to over 12 months achievement of weight loss corresponding to 10% of the initial weight in 12 months.
  It will be considered responder to therapy who reach such a result in 12 months

SECONDARY OUTCOMES:
body weight reduction by 5% compared to the initial weight | 6 months
  subjects will be considered responder to therapy if they reach such a result in 6 months , even if according Italian guidelines this will be considered failure
cardiovascular risk | 6, 12, 24 months
  cardiovascular risk according definition of Italian "Istituto Superiore di Sanità"
Attrition in the two groups | 6, 12, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Muggia, MD, Principal Investigator — Clinica Medica 2a
Locations (1):
- Clinica Medica 2A, Pavia, PV, Italy